CLINICAL TRIAL: NCT06037070
Title: Impact of Biological Factors on Dental Implant Osseointegration
Brief Title: Impact of Biological Factors on Dental Implant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Afya Sahib Diab Al-radha, Assistant Professor, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUOSU-202104
Record Dates: First submitted 2022-11-22; First posted 2023-09-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Dental Implant
Keywords: Dental implants; PRF; CBCT; osseointegration; bone density

STUDY DESIGN:
Intervention Model Description: Split-mouth trials
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group with PRF (Experimental): PRF placed inside the hole that prepared to place dental implant
  Interventions: Biological: Platelet Rich Fibrin
- control group (No Intervention): with out and additive

INTERVENTIONS:
Biological: Platelet Rich Fibrin — PRF will be injected inside the hole that prepared to place dental implant
  Arms: group with PRF

SUMMARY:
The goal of this randomized controlled trial is to compare the response of different bone densities to treatment with Platelet Rich Fibrin (PRF) in patients who need treatment with dental implant.

The main questions it aims to answer are:

* To investigate if bone reaction to PRF differ with different bone densities.
* To study the effect of PRF on dental implant healing and to assess its effectiveness in accelerating osseointegration.

Participants who need treatment with dental implant will be planned to include in this study and will be asked if they are willing to participate in this study voluntarily.

All the participants will be given an information sheet and a consent form which provides simple description about the present study and its importance to insure voluntary participation. The patients will be aware that they are completely free to withdraw from the research any time during the research time.

Platelet Rich Fibrin will be injected inside the hole that prepared to place dental implant in. Bone density will be evaluated, degree of osseointegration will be monitored.

DETAILED DESCRIPTION:
Materials and methods:

Two implants will be implanted at the same time, one will have PRF that will be injected inside the hole that prepared to place dental implant in [PRF is obtained from a blood sample is taken from the patient at the time of surgery in 10-mL tubes, the blood-containing tube is placed in a centrifuge at specially controlled rotations, temperature and time]. The other implant will not receive any treatment (the control one).

Evaluation of the results

* Evaluation of bone density in implant site will be determined using CBCT [ the same CBCT that have been used for planning dental implant treatment].

  ***[In dental implant treatment it is mandatory to perform CBCT for each patient, to ensure the accuracy of dental implant size and position, and to ensure there will be no damage to any vital structure during surgery (e.g. inferior dental nerve, maxillary sinus, …etc)].
* Evaluation of the degree of osseointegration will be performed using Osstell devise. [Osstell is a tool uses Resonance Frequency Analysis (RFA) that measures the frequency with which a device vibrates]. Measurement will be conducted at implant placement for a baseline reading and after 2weeks, 4weeks, 8 weeks, 10 weeks, 12 weeks.
* Evaluate pain by visual analogue score (VAS).
* Estimate of the complete blood picture, vit D, Ca and K will obtained from laboratory results.

ELIGIBILITY:
Inclusion criteria

* Non- smoker.
* No medical history of any systemic diseases that affect the bone metabolism.
* Did not receive any systemic drugs.
* Has edentulous area that needs at least two successive implants.

The exclusion criteria were as follows:

* Systemic disease or medication compromising bone and soft tissue healing.
* Pathology in the edentulous region.
* Bruxism.
* Disease of the oral mucosa.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
osseointegration | Immediately after surgery, after two weeks, 4 weeks, 6 weeks, 8weeks, 10 weeks, and 12 weeks
  Evaluation of the changes in the degree of osseointegration will be performed using Osstell devise.
Bone density | before surgery, with the treatment plan preparation
  Determined using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Afya SD Al-radha, Ph. D, Principal Investigator — College of Dentistry / Mustansiriyah University, P.O. Box: 14022,Baghdad, Iraq
Locations (1):
- Kadhimiya Teaching HospitalKadhimiya Educational Hospital, Baghdad, Alkadhmiya City, Iraq

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: after publication of the research, No end date.
Access Criteria: Anyone who wishes to access the data.
URL: http://myaccount.google.com/?utm_source=OGB&utm_medium=app&pli=1

DOCUMENTS (1):
  • Informed Consent Form (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT06037070/ICF_000.pdf